CLINICAL TRIAL: NCT01685281
Title: Randomized, Double-blind, Single-center, Dose-finding Study Designed to Compare Two Doses of MG01CI (Metadoxine Extended Release) and Placebo in Adults With Predominantly Inattentive Attention Deficit Hyperactivity Disorder
Brief Title: Study Comparing Two Doses of MG01CI and Placebo in Adults With Predominantly Inattentive Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AL011
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: ADHD Predominantly Inattentive Type
Keywords: ADHD , Inattention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — metadoxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metadoxine (MG01CI) 1400 mg (Active Comparator): single dose of Metadoxine (MG01CI) 1400 mg
  Interventions: Drug: Metadoxine (MG01CI)
- Metadoxine (MG01CI) 700 mg (Active Comparator): Single dose of Metadoxine (MG01CI) 700 mg
  Interventions: Drug: Metadoxine (MG01CI)
- Placebo (Placebo Comparator): Single dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metadoxine (MG01CI) — MG01CI is an orally administered extended release formulation of metadoxine. Doses: 1400 mg and 700 mg and Placebo
  Other Names: metadoxil
  Arms: Metadoxine (MG01CI) 1400 mg; Metadoxine (MG01CI) 700 mg
Drug: Placebo — Placebo tablets will be similar in appearance (color and size) to the investigational product
  Arms: Placebo

SUMMARY:
study objectives are to compare the efficacy, safety and tolerability of two doses of MG01CI (1400 mg and 700 mg) to Placebo for the treatment of symptoms in adults diagnosed with PI-ADHD.

subjects will be randomly assigned in a 1:1:1 ratio to one of three treatment sequences as follows:

1. week 1:1400 mg, week 2:700 mg, week 3:placebo
2. week 1:700 mg,week 2: placebo,week 3:1400 mg
3. week 1: placebo, week2:1400 mg, week 3 700 mg

The study will consist of three periods: a screening period of up to one week, a 3-week double-blind treatment period, and a one-week safety follow-up period.

DETAILED DESCRIPTION:
The purpose of this dose finding study is to compare two doses of MG01CI (1400 mg and 700 mg) to Placebo, in adult subjects with PI-ADHD. A crossover study design will allow evaluation of safety/tolerability and efficacy using validated computerized tests.

subjects will be randomly assigned in a 1:1:1 ratio to one of three treatment sequences as follows:

1. week 1:1400 mg, week 2:700 mg, week 3:placebo
2. week 1:700 mg,week 2: placebo,week 3:1400 mg
3. week 1: placebo, week2:1400 mg, week 3 700 mg

Overview of Study Visits

Screening Period:

Visit 1 - Screening/Baseline Visit (up to 7 days prior to dosing)

Treatment Period:

Visit 2 - Day 0 (Randomization Visit) Visit 3 - Day 7 ± 3 days Visit 4 - Day 14 ± 3 days Visit 5 - Day 21 ± 3 days

Follow-up period:

Visit 6 - Day 28 ± 3 days

Study duration for each subject will be up to 35 days .

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women, 18 to 55 years old
2. Diagnosed with predominantly inattentive ADHD based on DSM-IV criteria for ADHD as assessed by the Adult ADHD Clinician Diagnostic Scale (ACDS V1.2);
3. Clinical severity of at least a moderate level (Clinical Global Impression score of 4 or above)
4. TOVA ADHD score of -1.8 or below at Screening /Baseline
5. Women with childbearing potential must agree to use effective contraceptive and have negative urine pregnancy test at screening visit
6. Able to attend the clinic regularly and reliably
7. Able to swallow tablets/capsules
8. Able to understand, read, write and speak Hebrew fluently to complete study related materials
9. Able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

1. Subjects with ADHD not otherwise specified (NOS) diagnosis
2. Subjects with combined type or predominantly hyperactive impulsive ADHD diagnoses
3. Subjects with current Axis I diagnosis on SCID
4. Subjects with lifetime bipolar or psychosis
5. Subjects in treatment for Axis I disorders, even if the disorder is remitted
6. Subjects who were non-responders to at least two adequately administered ADHD treatments
7. Subjects with any medical or psychiatric condition common diseases such as hypertension, type 2 diabetes mellitus, hyperlipidemia, etc. are allowed per the Investigator's judgment, as long as they are stable and controlled by medical therapy that is constant for at least 8 weeks prior to randomization and throughout the study
8. Any prescription or non-prescription ADHD medications during the 14 days (for stimulants) or 28 days (for non-stimulants and other psychotropics) prior to the screening visit
9. Known or suspected HIV-positive or with advanced diseases such as AIDS, Hepatitis C, Hepatitis B or tuberculosis
10. History of allergy or sensitivity to B complex vitamins
11. History or suspicion of PDD, NLD or other psychotic conditions
12. Use of Vitamin B throughout the study (either alone or in any multi-vitamin)
13. Use of ADHD medications throughout the study
14. Use of any psychotropic medications throughout the study
15. Use of investigational medication/treatment in the past 30 days prior to the screening visit
16. Use of any medication or food supplement unless cleared by the medical monitor during the 14-day period before randomization
17. Current (or history within the last 6 months) of drug dependence or substance abuse disorder according to DSM-IV-TR criteria (excluding nicotine). Subjects should also agree to refrain from significantly changing consumption of caffeine during the study.
18. Suicidality, defined as active ideation, intent or plan, or any lifetime attempt (CSSRS)
19. Subjects who cannot complete any study instruments or questionnaires
20. Any relation to the Sponsor, Investigator or study staff
21. Any condition, which in the opinion of the Principal Investigator would place the subject at risk or influence the conduct of the study or interpretation of results, including (but not limited to) abnormally low intellectual capacity.
22. Subjects who cannot fully comprehend the implications of the protocol or comply with its requirements or are capable to follow the study schedule for any reason
23. Women of childbearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test and agree to use a reliable method of birth control (e.g., oral contraceptives or Norplant®; a reliable barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam]; intrauterine devices; partner with vasectomy; or abstinence) during the study. Note that this inclusion criterion applies only to females of childbearing potential. Females of childbearing potential are defined as women not surgically sterilized and between menarche and 2 years post-menopause

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in TOVA ADHD score from Screening/Baseline to 4 hours post-dose; | 4 weeks
  TOVA® is a computerized test that provides information about an individual's sustained attention, speed and consistency of responding, and behavioral self-regulation and executive functioning

SECONDARY OUTCOMES:
Change in CANTAB sub-scores from baseline (Visit 2) to 4 hours post-dose; | 4 weeks
  The CANTAB is a computerized test assessing the key cognitive deficits present in ADHD. Sub-scores will include spatial working memory (SWM), stop signal task (SST), rapid visual information processing (RVP), and reaction time (RTI).
Change in TOVA sub-scores from Screening/Baseline to 4 hours post-dose | 4 weeks
Number of participants who withdrew early from the study due to AE | 5 weeks

OTHER OUTCOMES:
Number of Adverse Events | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iris Manor, Dr., Principal Investigator — Geha Medical center
Locations (1):
- Geha Medical Centre, Petah Tikva, Israel

REFERENCES:
- [Derived] Manor I, Rubin J, Daniely Y, Adler LA. Attention benefits after a single dose of metadoxine extended release in adults with predominantly inattentive ADHD. Postgrad Med. 2014 Sep;126(5):7-16. doi: 10.3810/pgm.2014.09.2795. PMID 25295645